CLINICAL TRIAL: NCT01788228
Title: Safety and Tolerability of GSK 1557484A Vaccine in Adults at Occupational Risk for Influenza A (H5N1) Exposure
Brief Title: Safety and Tolerability Study of GlaxoSmithKline (GSK)1557484A Vaccine in Adults at Occupational Risk for Influenza A (H5N1) Exposure
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 116861
Record Dates: First submitted 2013-01-31; First posted 2013-02-11 (Estimated); Results first posted 2015-04-07 (Estimated); Last update posted 2020-06-23 (Actual); Status verified 2020-06

CONDITIONS: Influenza; Influenza Vaccines
Keywords: Vaccine; Occupational exposure; Influenza; H5N1
MeSH Terms: conditions — Influenza, Human

ARMS (2):
- Influenza A (H5N1) Virus monovalent vaccine 18-64 Years Group (Experimental): Subjects 18-64 years of age received 2 doses of Influenza A (H5N1) Virus Monovalent Vaccine, Adjuvanted (A/Indonesia) at Days 0 and 21. The vaccine was administered intramuscularly in the deltoid of the non-dominant arm at Day 0 and dominant arm at Day 21.
  Interventions: Biological: Influenza A (H5N1) Virus Monovalent Vaccine, Adjuvanted (A/Indonesia)
- Influenza A (H5N1) Virus monovalent vaccine > 64 Years Group (Experimental): Subjects >64 years of age received 2 doses of Influenza A (H5N1) Virus Monovalent Vaccine, Adjuvanted (A/Indonesia) at Days 0 and 21. The vaccine was administered intramuscularly in the deltoid of the non-dominant arm at Day 0 and dominant arm at Day 21.
  Interventions: Biological: Influenza A (H5N1) Virus Monovalent Vaccine, Adjuvanted (A/Indonesia)

INTERVENTIONS:
Biological: Influenza A (H5N1) Virus Monovalent Vaccine, Adjuvanted (A/Indonesia) — 2 doses administered intramuscularly (IM) in deltoid region of arm at the Day 0 and Day 21 visits.
  Other Names: GSK1557484A vaccine

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of GSK Biologicals' vaccine GSK1557484A against pandemic avian (H5N1) influenza in adults at occupational risk of exposure to the virus.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who, in the opinion of the investigator can and will comply with the requirements of the protocol.
* Male or female adults ≥18 years of age at time of first study vaccination.
* Written informed consent obtained from the subject.
* Subjects who are at risk of occupational exposure to H5N1 influenza viruses based on exposure, or potential exposure during either (a) laboratory operations with live H5N1 virus, (b) production of H5N1 vaccines, or (c) conduct of epidemiological investigations of H5N1 cases.
* Stable health status as defined by absence of a health event satisfying the definition of a serious adverse event, or a change in an ongoing drug therapy due to therapeutic failure or symptoms of drug toxicity, within 30 days prior to enrollment.
* Female subjects of non-childbearing potential may be enrolled in the study. Non-childbearing potential is defined as current tubal ligation, hysterectomy, ovariectomy or post-menopause.
* Female subjects of childbearing potential may be enrolled in the study, if they have practiced adequate contraception for 30 days prior to vaccination, and have a negative pregnancy test on the day of vaccination, and agree to practice adequate contraception for two months following the last dose of vaccine.

Exclusion Criteria:

* Presence or evidence of neurological or psychiatric diagnoses which, although stable, are deemed by the investigator to render the potential subject unable/unlikely to provide accurate safety reports.
* Presence of a temperature ≥ 38.0ºC (≥100.4ºF) or acute symptoms greater than "mild" severity on the scheduled date of first vaccination.

NOTE: The subject may be vaccinated at a later date, provided symptoms have resolved, vaccination occurs within the window specified by the protocol, and all other eligibility criteria continue to be satisfied.

* Significant risk of complications from intramuscular injections due to disorder of coagulation. Persons receiving prophylactic antiplatelet medications, e.g., low-dose aspirin, and without a clinically-apparent bleeding tendency, are eligible. Assessment of risk of injection complications should be made in the context of individual subject risk of H5N1 virus infection.
* An acute evolving neurological disorder or Guillain Barré Syndrome within 42 days of receipt of prior seasonal or pandemic influenza vaccine.
* Administration of an inactive vaccine within 14 days or of a live attenuated vaccine within 30 days before the first dose of study vaccine.
* Planned administration of any vaccine other than the study vaccine before Day 42.
* Any known or suspected allergy to any constituent of influenza vaccines or component used in the manufacturing process of the study vaccine including a history of anaphylactic-type reaction to consumption of eggs; or a history of severe adverse reaction to a previous influenza vaccine.
* Known pregnancy or a positive urine beta-human chorionic gonadotropin (β-hCG) test result before the first vaccination.
* Lactating or nursing women.
* Any condition which, in the opinion of the investigator, prevents the subject from participating in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2013-03-22 (Actual); Primary Completion 2014-03-27 (Actual); Study Completion 2015-02-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (3):
- United States (3):
  - GSK Investigational Site, Stockbridge, Georgia
  - GSK Investigational Site, Rockville, Maryland
  - GSK Investigational Site, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (click on the link provided below)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://www.clinicalstudydatarequest.com/SearchAllPostings.aspx?searchparam=116861

REFERENCES:
- [Background] Standaert B, Dort T, Linden J, Madan A, Bart S, Chu L, Hayney MS, Kosinski M, Kroll R, Malak J, Meier G, Segall N, Schuind A. Usability of daily SF36 questionnaires to capture the QALD variation experienced after vaccination with AS03A-adjuvanted monovalent influenza A (H5N1) vaccine in a safety and tolerability study. Health Qual Life Outcomes. 2019 May 6;17(1):80. doi: 10.1186/s12955-019-1147-4. PMID 31060567

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Influenza A (H5N1) Virus Monovalent Vaccine 18-64 Years Group | Influenza A (H5N1) Virus Monovalent Vaccine > 64 Years Group
Started | 49 | 1
Completed | 48 | 1
Not Completed | 1 | 0
Not completed — Migrated/moved from study area | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Influenza A (H5N1) Virus Monovalent Vaccine 18-64 Years Group | Influenza A (H5N1) Virus Monovalent Vaccine > 64 Years Group | Total
Number analyzed (Participants) | 49 | 1 | 50
Age, Continuous [Mean (Standard Deviation); unit: Years] | 42.5 (10.7) | 85.0 | 43.35 (12.18)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 0 | 28
  Male | 21 | 1 | 22

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Reporting Any and Grade 3 Solicited Local Symptoms Overall and by Age Category (18-64 and >64 Years of Age).
Description: Solicited local symptoms assessed were pain, redness and swelling. Any was defined as any solicited local symptom reported irrespective of intensity. Grade 3 pain was defined as significant pain at rest that prevented normal everyday activities. Grade 3 redness and swelling was greater than 100 millimeters (mm) i.e. >100mm.
Time Frame: During a 7-day follow-up period (Days 0-6) after each vaccination
Population: Analysis was performed on the Total Vaccinated cohort, which included all vaccinated subjects for whom safety data were available.
Measure: Count of Participants; unit: Participants
Groups:
- Influenza A (H5N1) Virus Monovalent Vaccine Group: Subjects ≥18 years of age received 2 doses of Influenza A (H5N1) Virus Monovalent Vaccine, Adjuvanted (A/Indonesia) at Days 0 and 21. The vaccine was administered intramuscularly in the deltoid of the nondominant armat Day 0 and dominant arm at Day 21.
Arm/Group | Influenza A (H5N1) Virus Monovalent Vaccine 18-64 Years Group | Influenza A (H5N1) Virus Monovalent Vaccine > 64 Years Group | Influenza A (H5N1) Virus Monovalent Vaccine Group
Number analyzed (Participants) | 49 | 1 | 50
Participants
  Any Pain | 45 | 1 | 46
  Grade 3 Pain | 4 | 0 | 4
  Any Redness | 6 | 0 | 6
  Grade 3 Redness | 0 | 0 | 0
  Any Swelling | 7 | 0 | 7
  Grade 3 Swelling | 0 | 0 | 0

2. Primary Outcome: Number of Subjects Reporting Any, Grade 3 and Related Solicited General Symptoms Overall and by Age Category (18-64 and >64 Years of Age).
Description: Solicited general symptoms assessed were fatigue, gastrointestinal symptoms, headache, joint pain, muscle ache, shivering, sweating and fever [oral temperature above 38.0 degrees Celsius (°C)]. Gastrointestinal symptoms included nausea, vomiting, diarrhea and/or abdominal pain. Any = any solicited general symptom reported irrespective of intensity and relationship to vaccination. Related = symptoms considered by the investigator to have a causal relationship to vaccination. Grade 3 symptoms = symptoms that prevented normal activity. Grade 3 fever = axillary temperature ≥ 39.0°C and ≤40°C.
Time Frame: During a 7-day follow-up period (Days 0-6) after each vaccination
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Influenza A (H5N1) Virus Monovalent Vaccine 18-64 Years Group | Influenza A (H5N1) Virus Monovalent Vaccine > 64 Years Group | Influenza A (H5N1) Virus Monovalent Vaccine Group
Number analyzed (Participants) | 49 | 1 | 50
Participants
  Any Fatigue | 27 | 0 | 27
  Grade 3 Fatigue | 1 | 0 | 1
  Related Fatigue | 26 | 0 | 26
  Any Gastrointestinal symptoms | 12 | 0 | 12
  Grade 3 Gastrointestinal symptoms | 2 | 0 | 2
  Related Gastrointestinal symptoms | 8 | 0 | 8
  Any Headache | 20 | 0 | 20
  Grade 3 Headache | 2 | 0 | 2
  Related Headache | 17 | 0 | 17
  Any Joint pain | 14 | 0 | 14
  Grade 3 Joint pain | 1 | 0 | 1
  Related Joint pain | 13 | 0 | 13
  Any Muscle ache | 33 | 0 | 33
  Grade 3 Muscle ache | 1 | 0 | 1
  Related Muscle ache | 31 | 0 | 31
  Any Shivering | 10 | 0 | 10
  Grade 3 Shivering | 1 | 0 | 1
  Related Shivering | 8 | 0 | 8
  Any Sweating | 7 | 0 | 7
  Grade 3 Sweating | 1 | 0 | 1
  Related Sweating | 5 | 0 | 5
  Any Fever (≥38°C) | 1 | 0 | 1
  Grade 3 Fever (≥39°C and ≤40°C) | 0 | 0 | 0
  Related Fever | 0 | 0 | 0

3. Primary Outcome: Number of Subjects Reporting Any Unsolicited AEs, Overall and by Age Category (18-64 and >64 Years of Age)
Description: Unsolicited AE covers any AE reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any was defined as occurrence of any unsolicited symptom regardless of intensity grade or relation to vaccination. Related was defined as an unsolicited symptom assessed as causally related to the study vaccination.
Time Frame: During the 21-day (Days 0-20 post dose 1 and Days 21-41 post dose 2) post-vaccination period
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Influenza A (H5N1) Virus Monovalent Vaccine 18-64 Years Group | Influenza A (H5N1) Virus Monovalent Vaccine > 64 Years Group | Influenza A (H5N1) Virus Monovalent Vaccine Group
Number analyzed (Participants) | 49 | 1 | 50
Participants
  Any unsolicited AEs | 10 | 0 | 10
  Related unsolicited AEs | 4 | 0 | 4

4. Secondary Outcome: Number of Subjects Reporting Any or Related Medically Attended Adverse Events (MAEs)
Description: MAEs refer to events that required medical attention defined as hospitalization, an emergency room visit or a visit to or from medical personnel (medical doctor) for any reason. Related = symptom assessed by the investigator as causally related to the study vaccination.
Time Frame: During the entire study period (Day 0 to Day 385)
Population: Analysis was performed on the Total Vaccinated cohort included all vaccinated subjects for whom safety data were available.
Measure: Count of Participants; unit: Participants
Arm/Group | Influenza A (H5N1) Virus Monovalent Vaccine 18-64 Years Group | Influenza A (H5N1) Virus Monovalent Vaccine > 64 Years Group
Number analyzed (Participants) | 49 | 1
Participants
  Any MAEs | 9 | 0
  Related MAEs | 0 | 0

5. Secondary Outcome: Number of Subjects Reporting Any and Related Potential Immune-Mediated Diseases (pIMDs)
Description: Potential immune-mediated diseases (pIMDs) were defined as a subset of adverse events (AEs) that included autoimmune diseases and other inflammatory and/or neurologic disorders of interest which may or may not have an autoimmune aetiology. Any was defined as occurrence of any pIMD regardless of intensity grade or relation to vaccination. Related was defined as pIMD(s) considered by the investigator to have a causal relationship to vaccination.
Time Frame: During the entire study period (Day 0 to Day 385)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Influenza A (H5N1) Virus Monovalent Vaccine 18-64 Years Group | Influenza A (H5N1) Virus Monovalent Vaccine > 64 Years Group
Number analyzed (Participants) | 49 | 1
Participants
  Any pIMDs | 0 | 0
  Related pIMDs | 0 | 0

6. Secondary Outcome: Number of Subjects Reporting Any and Related Serious Adverse Events (SAEs)
Description: A serious adverse event was any untoward medical occurrence that: resulted in death, was life-threatening, required hospitalization or prolongation of existing hospitalization, resulted in disability/incapacity or was a congenital anomaly/birth defect in the offspring of a study subject. Any was defined as occurrence of any symptom regardless of intensity grade or relation to vaccination and related was an event assessed by the investigator as causally related to the study vaccination.
Time Frame: During the entire study period (Day 0 to Day 385)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Influenza A (H5N1) Virus Monovalent Vaccine 18-64 Years Group | Influenza A (H5N1) Virus Monovalent Vaccine > 64 Years Group
Number analyzed (Participants) | 49 | 1
Participants
  Any SAEs | 0 | 0
  Related SAEs | 0 | 0

7. Secondary Outcome: Number of Subjects With Reported Adverse Pregnancy Outcomes
Description: Any = Occurrence of any adverse pregnancy outcomes regardless of intensity grade or relation to study vaccination. Related = Adverse pregnancy outcomes assessed by the investigator as causally related to the study vaccination
Time Frame: During the entire study period (Day 0 to Day 385)
Population: Analysis was performed on the Total Vaccinated cohort which included all vaccinated subjects for whom safety data were available.
Measure: Count of Participants; unit: Participants
Arm/Group | Influenza A (H5N1) Virus Monovalent Vaccine 18-64 Years Group | Influenza A (H5N1) Virus Monovalent Vaccine > 64 Years Group
Number analyzed (Participants) | 49 | 1
Participants
  Any adverse pregnancy outcome(s) | 0 | 0
  Related adverse pregnancy outcomes | 0 | 0

8. Secondary Outcome: Assessment of Changes From Baseline (Day 0) in the SF-36v2 Daily Questionnaire Subscale Component, Summary Component and QALY Scores
Description: The assessed parameters for change from baseline were Physical functioning (PF), Physical-health related role limitations (RP), Bodily pain (BP), General health (GH), Vitality (VT), Social functioning (SF), Emotional health related role limitations (RE), Mental health (MH) defined as subscale component, and physical (PCS) and mental (MCS) component defined as summary components, and Quality Adjusted Life Years (QALY). See methodology details in outcome 11 description. For all subscale components, scores range from 0 to 100, with high scores indicating high levels of functioning/quality of life. Subscale component scores are averaged to compute the summary component score and QALY score. Median and range of the change from baseline of the SF-36v2 score are presented for each component and time point. Analyses by age category were not performed for the daily SF-36v2 questionnaire results.
Time Frame: Day 0 (baseline) and at each day from Day 1 to Day 7 post first vaccine dose
Population: Analysis was performed on the Total Vaccinated cohort which included all vaccinated subjects. Only the subjects with available score test results were included.
Measure: Median (Full Range); unit: SF-36 daily score
Groups:
- Influenza A (H5N1) Virus Monovalent Vaccine Group: Subjects received 2 doses of Influenza A (H5N1) Virus Monovalent Vaccine, Adjuvanted (A/Indonesia) at Days 0 and 21. The vaccine was administered intramuscularly in the deltoid of the nondominant arm at Day 0 and dominant arm at Day 21.
Arm/Group | Influenza A (H5N1) Virus Monovalent Vaccine Group
Number analyzed (Participants) | 49
SF-36 daily score
  PF : Day 1: number analyzed (Participants) | 47
  PF : Day 1 | 0.0000 [-17.3500 to 28.9200]
  RP : Day 1: number analyzed (Participants) | 47
  RP : Day 1 | 0.0000 [-17.6100 to 8.81]
  BP : Day 1 | 0.0000 [-30.7900 to 10.2600]
  GH : Day 1 | -1.3200 [-16.7700 to 8.8200]
  VT : Day 1 | 0.0000 [-21.7700 to 21.7700]
  SF : Day 1 | 0.0000 [-19.7700 to 14.8200]
  RE : Day 1: number analyzed (Participants) | 47
  RE : Day 1 | 0.0000 [-7.6400 to 11.4500]
  MH : Day 1 | 0.0000 [-22.3000 to 14.8700]
  PCS : Day 1: number analyzed (Participants) | 47
  PCS : Day 1 | -1.0300 [-22.5200 to 14.8900]
  MCS : Day 1: number analyzed (Participants) | 47
  MCS : Day 1 | 0.0400 [-14.8500 to 10.7900]
  QALY score : Day 1: number analyzed (Participants) | 47
  QALY score : Day 1 | 0.0000 [-0.2660 to 0.2200]
  PF : Day 2 | 0.0000 [-19.2800 to 28.9200]
  RP : Day 2: number analyzed (Participants) | 48
  RP : Day 2 | 0.0000 [-26.4200 to 8.81]
  BP : Day 2: number analyzed (Participants) | 48
  BP : Day 2 | 0.0000 [-23.2900 to 10.2600]
  GH : Day 2 | 0.0000 [-12.3600 to 8.8200]
  VT : Day 2 | 0.0000 [-21.7700 to 21.7700]
  SF : Day 2 | 0.0000 [-29.6600 to 14.8200]
  RE : Day 2: number analyzed (Participants) | 48
  RE : Day 2 | 0.0000 [-22.9000 to 11.4500]
  MH : Day 2 | 0.0000 [-32.2100 to 9.9100]
  PCS : Day 2: number analyzed (Participants) | 48
  PCS : Day 2 | -0.5100 [-22.3100 to 14.7400]
  MCS : Day 2: number analyzed (Participants) | 48
  MCS : Day 2 | 0.4700 [-19.3500 to 7.3200]
  QALY score : Day 2: number analyzed (Participants) | 48
  QALY score : Day 2 | 0.0000 [-0.3570 to 0.2550]
  PF : Day 3: number analyzed (Participants) | 48
  PF : Day 3 | 0.0000 [-34.7100 to 28.9200]
  RP : Day 3: number analyzed (Participants) | 48
  RP : Day 3 | 0.0000 [-30.8200 to 8.81]
  BP : Day 3: number analyzed (Participants) | 48
  BP : Day 3 | 0.0000 [-30.7900 to 15.0000]
  GH : Day 3 | 0.0000 [-13.2400 to 8.8200]
  VT : Day 3: number analyzed (Participants) | 48
  VT : Day 3 | 0.0000 [-19.0600 to 13.6100]
  SF : Day 3 | 0.0000 [-29.6600 to 19.7600]
  RE : Day 3: number analyzed (Participants) | 48
  RE : Day 3 | 0.0000 [-7.6400 to 11.4500]
  MH : Day 3: number analyzed (Participants) | 48
  MH : Day 3 | 0.0000 [-9.9100 to 7.4300]
  PCS : Day 3: number analyzed (Participants) | 47
  PCS : Day 3 | 0.0800 [-38.6400 to 13.3300]
  MCS : Day 3: number analyzed (Participants) | 47
  MCS : Day 3 | 0.6200 [-9.1700 to 9.7200]
  QALY score : Day 3: number analyzed (Participants) | 47
  QALY score : Day 3 | 0.0000 [-0.4030 to 0.2490]
  PF : Day 4: number analyzed (Participants) | 48
  PF : Day 4 | 0.0000 [-34.7100 to 28.9200]
  RP : Day 4: number analyzed (Participants) | 48
  RP : Day 4 | 0.0000 [-35.2300 to 8.81]
  BP : Day 4: number analyzed (Participants) | 48
  BP : Day 4 | 0.0000 [-30.7900 to 11.0500]
  GH : Day 4 | 0.0000 [-13.2400 to 8.8200]
  VT : Day 4 | 0.0000 [-21.7700 to 21.7700]
  SF : Day 4 | 0.0000 [-29.6600 to 19.7600]
  RE : Day 4: number analyzed (Participants) | 48
  RE : Day 4 | 0.0000 [-30.5400 to 11.4500]
  MH : Day 4 | 0.0000 [-12.3900 to 7.4300]
  PCS : Day 4: number analyzed (Participants) | 47
  PCS : Day 4 | 0.0000 [-33.6200 to 14.0400]
  MCS : Day 4: number analyzed (Participants) | 48
  MCS : Day 4 | 0.0750 [-13.2200 to 9.7200]
  QALY score : Day 4: number analyzed (Participants) | 47
  QALY score : Day 4 | 0.0000 [-0.4030 to 0.2910]
  PF : Day 5 | 0.0000 [-34.7100 to 28.9200]
  RP : Day 5 | 0.0000 [-33.0300 to 8.81]
  BP : Day 5 | 0.0000 [-30.7900 to 15.0000]
  GH : Day 5 | 0.0000 [-17.6400 to 8.8200]
  VT : Day 5 | 0.0000 [-21.7700 to 21.7700]
  SF : Day 5 | 0.0000 [-24.7100 to 19.7600]
  RE : Day 5 | 0.0000 [-38.1700 to 11.4500]
  MH : Day 5 | 0.0000 [-14.8600 to 12.3900]
  PCS : Day 5 | 0.0700 [-31.2600 to 14.0400]
  MCS : Day 5 | 0.6000 [-14.2000 to 14.0500]
  QALY score : Day 5: number analyzed (Participants) | 48
  QALY score : Day 5 | 0.0000 [-0.3900 to 0.2910]
  PF : Day 6 | 0.0000 [-21.2100 to 28.9200]
  RP : Day 6 | 0.0000 [-17.6100 to 8.81]
  BP : Day 6 | 0.0000 [-23.2900 to 15.0000]
  GH : Day 6 | 0.0000 [-12.3600 to 8.8200]
  VT : Day 6 | 0.0000 [-24.4900 to 21.7700]
  SF : Day 6 | 0.0000 [-9.8900 to 19.7600]
  RE : Day 6 | 0.0000 [-19.0900 to 11.4500]
  MH : Day 6 | 0.0000 [-12.3900 to 7.4300]
  PCS : Day 6 | 0.0800 [-20.5900 to 14.0400]
  MCS : Day 6 | 0.4000 [-8.0600 to 9.7200]
  QALY score : Day 6 | 0.0000 [-0.3420 to 0.2910]
  PF : Day 7 | 0.0000 [-7.7100 to 28.9200]
  RP : Day 7 | 0.0000 [-19.8200 to 8.8100]
  BP : Day 7: number analyzed (Participants) | 48
  BP : Day 7 | 0.0000 [-15.0000 to 19.3400]
  GH : Day 7 | 0.0000 [-11.0300 to 8.8200]
  VT : Day 7: number analyzed (Participants) | 48
  VT : Day 7 | 0.0000 [-24.4900 to 10.8900]
  SF : Day 7 | 0.0000 [-4.9500 to 24.7100]
  RE : Day 7 | 0.0000 [-15.2700 to 11.4500]
  MH : Day 7: number analyzed (Participants) | 48
  MH : Day 7 | 0.0000 [-19.8200 to 7.4300]
  PCS : Day 7: number analyzed (Participants) | 48
  PCS : Day 7 | 0.1150 [-13.3900 to 14.0400]
  MCS : Day 7: number analyzed (Participants) | 48
  MCS : Day 7 | 0.3850 [-9.2200 to 9.7000]
  QALY score : Day 7: number analyzed (Participants) | 48
  QALY score : Day 7 | 0.0000 [-0.2230 to 0.2910]

9. Secondary Outcome: Assessment of Changes From Baseline (Day 0) in the SF-36v2 Weekly Health 8-score
Description: The assessed parameters for change from baseline were Physical functioning (PF), Physical-health related role limitations (RP), Bodily pain (BP), General health (GH), Vitality (VT), Social functioning (SF), Emotional health related role limitations (RE), Mental health (MH) defined as subscale component. For all subscale components, scores range from 0 to 100, with high scores indicating high levels of functioning/quality of life. Median and range of the change from baseline of the SF-36 score are presented for each component and time point. Analysis was carried out for all subjects regardless of age stratum.
Time Frame: Day 0 (baseline) and at Days 7 and 21 QoL evaluation (post dose 1) and Day 28 QoL evaluation (post dose 2)
Population: as for outcome 8
Measure: Median (Full Range); unit: SF-36 Weekly score
Groups:
- Influenza A (H5N1) Virus Monovalent Vaccine Group: Subjects received 2 doses of Influenza A (H5N1) Virus Monovalent Vaccine, Adjuvanted (A/Indonesia) at Days 0 and 21. The vaccine was administered intramuscularly in the deltoid of the non-dominant arm at Day 0 and dominant arm at Day 21.
Arm/Group | Influenza A (H5N1) Virus Monovalent Vaccine Group
Number analyzed (Participants) | 50
SF-36 Weekly score
  PF : Day 7: number analyzed (Participants) | 49
  PF : Day 7 | 0.000 [-1.93 to 28.92]
  PF : Day 21: number analyzed (Participants) | 48
  PF : Day 21 | 0.000 [-7.71 to 28.92]
  PF : Day 28: number analyzed (Participants) | 49
  PF : Day 28 | 0.000 [-5.78 to 28.92]
  RP: Day 7 | 0.000 [-17.61 to 8.81]
  RP: Day 21: number analyzed (Participants) | 49
  RP: Day 21 | 0.000 [-15.41 to 8.81]
  RP: Day 28 | 0.000 [-17.61 to 8.81]
  BP: Day 7: number analyzed (Participants) | 49
  BP: Day 7 | 0.000 [-26.85 to 19.34]
  BP: Day 21: number analyzed (Participants) | 48
  BP: Day 21 | 0.000 [-15.00 to 23.29]
  BP: Day 28: number analyzed (Participants) | 49
  BP: Day 28 | 0.000 [-11.05 to 15.00]
  GH: Day 7 | 0.000 [-9.93 to 7.50]
  GH: Day 21: number analyzed (Participants) | 49
  GH: Day 21 | 0.000 [-15.44 to 7.50]
  GH: Day 28 | 0.000 [-15.44 to 8.82]
  VT: Day 7 | 0.000 [-21.77 to 19.05]
  VT: Day 21: number analyzed (Participants) | 49
  VT: Day 21 | 2.720 [-10.89 to 13.61]
  VT: Day 28 | 0.000 [-13.61 to 16.33]
  SF: Day 7: number analyzed (Participants) | 49
  SF: Day 7 | 0.000 [-19.77 to 14.83]
  SF: Day 21: number analyzed (Participants) | 48
  SF: Day 21 | 0.000 [-9.89 to 9.89]
  SF: Day 28: number analyzed (Participants) | 49
  SF: Day 28 | 0.000 [-19.77 to 14.83]
  RE: Day 7 | 0.000 [-22.90 to 11.45]
  RE: Day 21: number analyzed (Participants) | 49
  RE: Day 21 | 0.000 [-22.90 to 11.45]
  RE: Day 28 | 0.000 [-11.45 to 11.45]
  MH: Day 7 | 0.000 [-14.87 to 7.43]
  MH: Day 21: number analyzed (Participants) | 49
  MH: Day 21 | 0.000 [-9.91 to 7.44]
  MH: Day 28 | 0.000 [-17.35 to 7.44]

10. Secondary Outcome: Assessment of Changes From Baseline (Day 0) in the SF-36v2 Weekly Questionnaire General Health Scores (Physical and Mental)
Description: The assessed parameters for change from baseline were physical and mental component defined as summary components (PCS and MCS) or general health scores (GHS). For all subscale component, scores range from 0 to 100, with high scores indicating high levels of functioning/quality of life. Subscale component scores are averaged to compute the summary component score. Median and range of the change from baseline of the SF-36v2 score are presented for each summary component and time point. Analysis was carried out for all subjects regardless of age stratum.
Time Frame: Day 0 (baseline) and at Days 7 and 21 QoL evaluation (post dose 1) and Day 28 QoL evaluation (post dose 2)
Population: as for outcome 8
Measure: Median (Full Range); unit: SF-36 weekly score
Arm/Group | Influenza A (H5N1) Virus Monovalent Vaccine Group
Number analyzed (Participants) | 49
SF-36 weekly score
  PCS, Day 7 | 0.000 [-11.19 to 13.58]
  PCS, Day 21: number analyzed (Participants) | 48
  PCS, Day 21 | 0.180 [-11.32 to 13.58]
  PCS, Day 28 | -0.290 [-6.36 to 13.58]
  MCS, Day 7 | 0.420 [-11.08 to 11.83]
  MCS, Day 21: number analyzed (Participants) | 48
  MCS, Day 21 | 0.095 [-5.10 to 7.33]
  MCS, Day 28 | 0.000 [-7.29 to 11.83]

11. Secondary Outcome: Assessment of Changes From Baseline (Day 0) for Quality Adjusted Life Years (QALY) Weekly Scores
Description: The assessed parameters for change from baseline were QALY scores. The methodology used for the analysis of the SF-36v2 questionnaire was detailed in Ware et al [Ware 2008]. The QualityMetric Health Outcomes Scoring Software was used to generate a Quality of Life analysis dataset based on the SF-36 questionnaire. QoL data were transformed to generate Quality-Adjusted Life Years (QALY) scores. A standard algorithm was developed for processing subjects' answers and producing QALY scores. For all subscale components, scores range from 0 to 100, with high scores indicating high levels of functioning/quality of life. Median and range of the change from baseline of the SF-36v2 score are presented for each time point. Analysis was carried out for all subjects regardless of age stratum.
Time Frame: Day 0 (baseline) and at Days 7 and 21 QoL evaluation (post dose 1) and Day 28 QoL evaluation (post dose 2)
Population: as for outcome 8
Measure: Median (Full Range); unit: SF-36 Weekly score
Arm/Group | Influenza A (H5N1) Virus Monovalent Vaccine Group
Number analyzed (Participants) | 48
SF-36 Weekly score
  QALY score : Day 7 | 0.000 [-0.25 to 0.33]
  QALY score : Day 21 | 0.000 [-0.25 to 0.33]
  QALY score : Day 28 | 0.000 [-0.19 to 0.33]

12. Secondary Outcome: Assessment of Changes From Baseline (Day 0) in the SF-36v2 Daily Questionnaire Subscale Component, Summary Component and QALY Scores for Subjects Who Reported at Least One Local or General Solicited AE Post First Vaccination.
Description: The assessed parameters for change from baseline were Physical functioning (PF), Physical-health related role limitations (RP), Bodily pain (BP), General health (GH), Vitality (VT), Social functioning (SF), Emotional health related role limitations (RE), Mental health (MH) defined as subscale component, and physical (PCS) and mental (MCS) component defined as summary components, and Quality Adjusted Life Years (QALY). For all subscale component, scores range from 0 to 100, with high scores indicating high levels of functioning/quality of life. Subscale component scores are averaged to compute the summary component score and QALY score. Median and range of the change from baseline of the SF-36v2 score are presented for each component and time point. Analyses by age category were not performed for the daily SF-36v2 questionnaire results.
Time Frame: Day 0 (baseline) and at each day from Day 1 to Day 7 post first vaccine dose
Population: Analysis was performed on the Total Vaccinated cohort which included all vaccinated subjects who reported at least one local or general solicited AE post first vaccination. Only the subjects with available score test results were included.
Measure: Median (Full Range); unit: SF-36 daily score
Arm/Group | Influenza A (H5N1) Virus Monovalent Vaccine Group
Number analyzed (Participants) | 47
SF-36 daily score
  PF : Day 1: number analyzed (Participants) | 45
  PF : Day 1 | 0.0000 [-17.3500 to 28.9200]
  RP : Day 1: number analyzed (Participants) | 45
  RP : Day 1 | 0.0000 [-17.6100 to 8.81]
  BP : Day 1 | -0.7900 [-30.7900 to 8.6800]
  GH : Day 1 | -1.3200 [-16.7700 to 8.8200]
  VT : Day 1 | 0.0000 [-21.7700 to 21.7700]
  SF : Day 1 | 0.0000 [-19.7700 to 14.8200]
  RE : Day 1: number analyzed (Participants) | 45
  RE : Day 1 | 0.0000 [-7.6400 to 11.4500]
  MH : Day 1 | 0.0000 [-22.3000 to 14.8700]
  PCS : Day 1: number analyzed (Participants) | 45
  PCS : Day 1 | -1.1000 [-22.5200 to 14.8900]
  MCS : Day 1: number analyzed (Participants) | 45
  MCS : Day 1 | 0.0400 [-14.8500 to 10.7900]
  QALY score : Day 1: number analyzed (Participants) | 45
  QALY score : Day 1 | 0.0000 [-0.2660 to 0.2200]
  PF : Day 2 | 0.0000 [-19.2800 to 28.9200]
  RP : Day 2: number analyzed (Participants) | 46
  RP : Day 2 | 0.0000 [-26.4200 to 8.81]
  BP : Day 2: number analyzed (Participants) | 46
  BP : Day 2 | 0.0000 [-23.2900 to 10.2600]
  GH : Day 2 | 0.0000 [-12.3600 to 8.8200]
  VT : Day 2 | 0.0000 [-21.7700 to 21.7700]
  SF : Day 2 | 0.0000 [-29.6600 to 14.8200]
  RE : Day 2: number analyzed (Participants) | 46
  RE : Day 2 | 0.0000 [-22.9000 to 11.4500]
  MH : Day 2 | 0.0000 [-32.2100 to 4.9600]
  PCS : Day 2: number analyzed (Participants) | 46
  PCS : Day 2 | -0.5500 [-22.3100 to 14.7400]
  MCS : Day 2: number analyzed (Participants) | 46
  MCS : Day 2 | 0.3950 [-19.3500 to 7.3200]
  QALY score : Day 2: number analyzed (Participants) | 46
  QALY score : Day 2 | 0.0000 [-0.3570 to 0.2550]
  PF : Day 3: number analyzed (Participants) | 46
  PF : Day 3 | 0.0000 [-34.7100 to 28.9200]
  RP : Day 3: number analyzed (Participants) | 46
  RP : Day 3 | 0.0000 [-30.8200 to 8.81]
  BP : Day 3: number analyzed (Participants) | 46
  BP : Day 3 | 0.0000 [-30.7900 to 15.0000]
  GH : Day 3 | 0.0000 [-13.2400 to 8.8200]
  VT : Day 3: number analyzed (Participants) | 46
  VT : Day 3 | 0.0000 [-19.0600 to 13.6100]
  SF : Day 3 | 0.0000 [-29.6600 to 19.7600]
  RE : Day 3: number analyzed (Participants) | 46
  RE : Day 3 | 0.0000 [-7.6400 to 11.4500]
  MH : Day 3: number analyzed (Participants) | 46
  MH : Day 3 | 0.0000 [-9.9100 to 7.4300]
  PCS : Day 3: number analyzed (Participants) | 45
  PCS : Day 3 | 0.0800 [-38.6400 to 13.3300]
  MCS : Day 3: number analyzed (Participants) | 45
  MCS : Day 3 | 0.6000 [-9.1700 to 9.7200]
  QALY score : Day 3: number analyzed (Participants) | 45
  QALY score : Day 3 | 0.0000 [-0.4030 to 0.2490]
  PF : Day 4: number analyzed (Participants) | 46
  PF : Day 4 | 0.0000 [-34.7100 to 28.9200]
  RP : Day 4 | 0.0000 [-35.2300 to 8.81]
  BP : Day 4 | 0.0000 [-30.7900 to 11.0500]
  GH : Day 4 | 0.0000 [-13.2400 to 8.8200]
  VT : Day 4 | 0.0000 [-21.7700 to 21.7700]
  SF : Day 4 | 0.0000 [-29.6600 to 19.7600]
  RE : Day 4 | 0.0000 [-30.5400 to 11.4500]
  MH : Day 4 | 0.0000 [-12.3900 to 7.4300]
  PCS : Day 4: number analyzed (Participants) | 46
  PCS : Day 4 | 0.0350 [-33.6200 to 14.0400]
  MCS : Day 4 | 0.0600 [-13.2200 to 9.7200]
  QALY score : Day 4: number analyzed (Participants) | 46
  QALY score : Day 4 | 0.0000 [-0.4030 to 0.2910]
  PF : Day 5 | 0.0000 [-34.7100 to 28.9200]
  RP : Day 5 | 0.0000 [-33.0300 to 8.81]
  BP : Day 5 | 0.0000 [-30.7900 to 15.0000]
  GH : Day 5 | 0.0000 [-17.6400 to 8.8200]
  VT : Day 5 | 0.0000 [-21.7700 to 21.7700]
  SF : Day 5 | 0.0000 [-24.7100 to 19.7600]
  RE : Day 5 | 0.0000 [-38.1700 to 11.4500]
  MH : Day 5 | 0.0000 [-14.8600 to 12.3900]
  PCS : Day 5 | 0.0700 [-31.2600 to 14.0400]
  MCS : Day 5 | 0.3800 [-14.2000 to 14.0500]
  QALY score : Day 5: number analyzed (Participants) | 46
  QALY score : Day 5 | 0.0000 [-0.3900 to 0.2910]
  PF : Day 6 | 0.0000 [-21.2100 to 28.9200]
  RP : Day 6 | 0.0000 [-17.6100 to 8.81]
  BP : Day 6 | 0.0000 [-23.2900 to 15.0000]
  GH : Day 6 | 0.0000 [-12.3600 to 8.8200]
  VT : Day 6 | 0.0000 [-24.4900 to 21.7700]
  SF : Day 6 | 0.0000 [-9.8900 to 19.7600]
  RE : Day 6 | 0.0000 [-19.0900 to 11.4500]
  MH : Day 6 | 0.0000 [-12.3900 to 7.4300]
  PCS : Day 6 | 0.0800 [-20.5900 to 14.0400]
  MCS : Day 6 | 0.0700 [-8.0600 to 9.7200]
  QALY score : Day 6 | 0.0000 [-0.3420 to 0.2910]
  PF : Day 7 | 0.0000 [-7.7100 to 28.9200]
  RP : Day 7 | 0.0000 [-19.8200 to 8.8100]
  BP : Day 7: number analyzed (Participants) | 46
  BP : Day 7 | 0.0000 [-15.0000 to 19.3400]
  GH : Day 7 | 0.0000 [-11.0200 to 8.8200]
  VT : Day 7: number analyzed (Participants) | 46
  VT : Day 7 | 0.0000 [-24.4900 to 10.8900]
  SF : Day 7 | 0.0000 [-4.9500 to 24.7100]
  RE : Day 7 | 0.0000 [-15.2700 to 11.4500]
  MH : Day 7: number analyzed (Participants) | 46
  MH : Day 7 | 0.0000 [-19.8200 to 7.4300]
  PCS : Day 7: number analyzed (Participants) | 46
  PCS : Day 7 | 0.1150 [-13.3900 to 14.0400]
  MCS : Day 7: number analyzed (Participants) | 46
  MCS : Day 7 | 0.2100 [-9.2200 to 9.7000]
  QALY score : Day 7: number analyzed (Participants) | 46
  QALY score : Day 7 | 0.0000 [-0.2230 to 0.2910]

13. Secondary Outcome: Assessment of Changes From Baseline (Day 0) for the SF-36v2 Weekly Health 8-score for All Subjects Who Did and Who Did Not Report Any Grade 3 Solicited Symptoms Post Vaccination.
Description: Median and range of the change from baseline of the SF-36v2 score are presented for each component and time point. The assessed parameters for change from baseline were Physical functioning (PF), Physical-health related role limitations (RP), Bodily pain (BP), General health (GH), Vitality (VT), Social functioning (SF), Emotional health related role limitations (RE), Mental health (MH) defined as subscale component. For all subscale component, scores range from 0 to 100, with high scores indicating high levels of functioning/quality of life. There was only 1 study participant > 64 years of age and that experienced no grade 3 solicited symptoms. Hence, weekly questionnaire was assessed only on the 18-64 age category subjects.
Time Frame: Day 0 (baseline) and at Days 7 and 21 QoL evaluation (post dose 1) and Day 28 QoL evaluation (post dose 2)
Population: Analysis was performed on the Total Vaccinated cohort (18-64 years of age) which included all vaccinated subjects within 18 to 64 years of age and for whom safety data were available. Only subjects with available score test results were included.
Measure: Median (Full Range); unit: SF-36 Weekly score
Arm/Group | Influenza A (H5N1) Virus Monovalent Vaccine 18-64 Years Group
Number analyzed (Participants) | 49
SF-36 Weekly score
  PF, Grade 3 AE, Day 7: number analyzed (Participants) | 6
  PF, Grade 3 AE, Day 7 | 0.000 [0.00 to 0.00]
  PF, Grade 3 AE, Day 21: number analyzed (Participants) | 6
  PF, Grade 3 AE, Day 21 | 0.000 [0.00 to 0.00]
  PF, Grade 3 AE, Day 28: number analyzed (Participants) | 6
  PF, Grade 3 AE, Day 28 | 0.000 [-5.78 to 0.00]
  RP, Grade 3 AE, Day 7: number analyzed (Participants) | 6
  RP, Grade 3 AE, Day 7 | 0.000 [-17.61 to 0.00]
  RP, Grade 3 AE, Day 21: number analyzed (Participants) | 6
  RP, Grade 3 AE, Day 21 | 0.000 [0.00 to 0.00]
  RP, Grade 3 AE, Day 28: number analyzed (Participants) | 6
  RP, Grade 3 AE, Day 28 | 0.000 [-15.41 to 0.00]
  BP, Grade 3 AE, Day 7: number analyzed (Participants) | 6
  BP, Grade 3 AE, Day 7 | 0.000 [-10.26 to 8.29]
  BP, Grade 3 AE, Day 21: number analyzed (Participants) | 6
  BP, Grade 3 AE, Day 21 | 0.000 [-10.26 to 23.29]
  BP, Grade 3 AE, Day 28: number analyzed (Participants) | 6
  BP, Grade 3 AE, Day 28 | 0.000 [-6.32 to 6.32]
  GH, Grade 3 AE, Day 7: number analyzed (Participants) | 6
  GH, Grade 3 AE, Day 7 | 0.215 [-2.21 to 7.50]
  GH, Grade 3 AE, Day 21: number analyzed (Participants) | 6
  GH, Grade 3 AE, Day 21 | 0.660 [-2.21 to 7.50]
  GH, Grade 3 AE, Day 28: number analyzed (Participants) | 6
  GH, Grade 3 AE, Day 28 | 0.215 [-2.21 to 8.82]
  VT, Grade 3 AE, Day 7: number analyzed (Participants) | 6
  VT, Grade 3 AE, Day 7 | 0.000 [-9.97 to 5.44]
  VT, Grade 3 AE, Day 21: number analyzed (Participants) | 6
  VT, Grade 3 AE, Day 21 | 1.365 [-5.44 to 5.44]
  VT, Grade 3 AE, Day 28: number analyzed (Participants) | 6
  VT, Grade 3 AE, Day 28 | 1.360 [-2.72 to 5.44]
  SF, Grade 3 AE, Day 7: number analyzed (Participants) | 6
  SF, Grade 3 AE, Day 7 | -4.945 [-19.77 to 0.00]
  SF, Grade 3 AE, Day 21: number analyzed (Participants) | 6
  SF, Grade 3 AE, Day 21 | 0.000 [-9.89 to 0.00]
  SF, Grade 3 AE, Day 28: number analyzed (Participants) | 6
  SF, Grade 3 AE, Day 28 | 0.000 [-14.83 to 0.00]
  RE, Grade 3 AE, Day 7: number analyzed (Participants) | 6
  RE, Grade 3 AE, Day 7 | 0.000 [-15.27 to 0.00]
  RE, Grade 3 AE, Day 21: number analyzed (Participants) | 6
  RE, Grade 3 AE, Day 21 | 0.000 [0.00 to 0.00]
  RE, Grade 3 AE, Day 28: number analyzed (Participants) | 6
  RE, Grade 3 AE, Day 28 | 0.000 [-11.45 to 0.00]
  MH, Grade 3 AE, Day 7: number analyzed (Participants) | 6
  MH, Grade 3 AE, Day 7 | 1.235 [-2.48 to 2.47]
  MH, Grade 3 AE, Day 21: number analyzed (Participants) | 6
  MH, Grade 3 AE, Day 21 | 1.235 [-2.48 to 2.47]
  MH, Grade 3 AE, Day 28: number analyzed (Participants) | 6
  MH, Grade 3 AE, Day 28 | 1.235 [-2.48 to 2.47]
  PF, No Grade 3 AE, Day 7: number analyzed (Participants) | 42
  PF, No Grade 3 AE, Day 7 | 0.000 [-1.93 to 28.92]
  PF, No Grade 3 AE, Day 21: number analyzed (Participants) | 42
  PF, No Grade 3 AE, Day 21 | 0.000 [-7.71 to 28.92]
  PF, No Grade 3 AE, Day 28: number analyzed (Participants) | 42
  PF, No Grade 3 AE, Day 28 | 0.000 [-1.93 to 28.92]
  RP, No Grade 3 AE, Day 7: number analyzed (Participants) | 43
  RP, No Grade 3 AE, Day 7 | 0.000 [-15.41 to 8.81]
  RP, No Grade 3 AE, Day 21: number analyzed (Participants) | 43
  RP, No Grade 3 AE, Day 21 | 0.000 [-15.41 to 8.81]
  RP, No Grade 3 AE, Day 28: number analyzed (Participants) | 43
  RP, No Grade 3 AE, Day 28 | 0.000 [-17.61 to 8.81]
  BP, No Grade 3 AE, Day 7: number analyzed (Participants) | 42
  BP, No Grade 3 AE, Day 7 | 0.000 [-26.85 to 19.34]
  BP, No Grade 3 AE, Day 21: number analyzed (Participants) | 42
  BP, No Grade 3 AE, Day 21 | 0.000 [-15.00 to 15.00]
  BP, No Grade 3 AE, Day 28: number analyzed (Participants) | 42
  BP, No Grade 3 AE, Day 28 | 0.000 [-11.05 to 15.00]
  GH, No Grade 3 AE, Day 7: number analyzed (Participants) | 43
  GH, No Grade 3 AE, Day 7 | 0.000 [-9.93 to 6.61]
  GH, No Grade 3 AE, Day 21: number analyzed (Participants) | 43
  GH, No Grade 3 AE, Day 21 | 0.000 [-15.44 to 6.61]
  GH, No Grade 3 AE, Day 28: number analyzed (Participants) | 43
  GH, No Grade 3 AE, Day 28 | 0.000 [-15.44 to 6.62]
  VT, No Grade 3 AE, Day 7: number analyzed (Participants) | 43
  VT, No Grade 3 AE, Day 7 | 0.000 [-21.77 to 19.05]
  VT, No Grade 3 AE, Day 21: number analyzed (Participants) | 43
  VT, No Grade 3 AE, Day 21 | 2.720 [-10.89 to 13.61]
  VT, No Grade 3 AE, Day 28: number analyzed (Participants) | 43
  VT, No Grade 3 AE, Day 28 | 0.000 [-13.61 to 16.33]
  SF, No Grade 3 AE, Day 7: number analyzed (Participants) | 42
  SF, No Grade 3 AE, Day 7 | 0.000 [-19.77 to 14.83]
  SF, No Grade 3 AE, Day 21: number analyzed (Participants) | 42
  SF, No Grade 3 AE, Day 21 | 0.000 [-9.89 to 9.89]
  SF, No Grade 3 AE, Day 28: number analyzed (Participants) | 42
  SF, No Grade 3 AE, Day 28 | 0.000 [-19.77 to 14.83]
  RE, No Grade 3 AE, Day 7: number analyzed (Participants) | 43
  RE, No Grade 3 AE, Day 7 | 0.000 [-22.90 to 11.45]
  RE, No Grade 3 AE, Day 21: number analyzed (Participants) | 43
  RE, No Grade 3 AE, Day 21 | 0.000 [-22.90 to 11.45]
  RE, No Grade 3 AE, Day 28: number analyzed (Participants) | 43
  RE, No Grade 3 AE, Day 28 | 0.000 [-7.64 to 11.45]
  MH, No Grade 3 AE, Day 7: number analyzed (Participants) | 43
  MH, No Grade 3 AE, Day 7 | 0.000 [-14.87 to 7.43]
  MH, No Grade 3 AE, Day 21: number analyzed (Participants) | 43
  MH, No Grade 3 AE, Day 21 | 0.000 [-9.91 to 7.44]
  MH, No Grade 3 AE, Day 28: number analyzed (Participants) | 43
  MH, No Grade 3 AE, Day 28 | 0.000 [-17.35 to 7.44]

14. Secondary Outcome: Assessment of Changes From Baseline (Day 0) in the SF-36v2 Weekly Questionnaire General Health Scores(Physical and Mental) for Subjects Who Did and Who Did Not Report Any Grade 3 Solicited Symptoms Post Vaccination.
Description: Median and range of the change from baseline of the SF-36v2 score are presented for each component and time point. The assessed parameters for change from baseline were physical and mental component defined as summary components (PCS and MCS) or general health scores (GHS). For all subscale component, scores range from 0 to 100, with high scores indicating high levels of functioning/quality of life. Subscale component scores are averaged to compute the summary component score. There was only 1 study participant > 64 years of age and that experienced no grade 3 solicited symptoms. Hence, weekly questionnaire was assessed only on the 18-64 age category subjects.
Time Frame: Day 0 (baseline) and at Days 7 and 21 QoL evaluation (post dose 1) and Day 28 QoL evaluation (post dose 2)
Population: Analysis was performed on the Total Vaccinated cohort (18-64 years of age) which included all vaccinated subjects within 18 to 64 years of age and for whom safety data were available. Only the subjects with available score test results were included.
Measure: Median (Full Range); unit: SF-36 weekly score
Arm/Group | Influenza A (H5N1) Virus Monovalent Vaccine 18-64 Years Group
Number analyzed (Participants) | 48
SF-36 weekly score
  PCS, Grade 3 solicited AE (Day 7): number analyzed (Participants) | 6
  PCS, Grade 3 solicited AE (Day 7) | -0.370 [-7.20 to 2.49]
  PCS, Grade 3 solicited AE (Day 21): number analyzed (Participants) | 6
  PCS, Grade 3 solicited AE (Day 21) | 1.170 [-3.73 to 6.34]
  PCS, Grade 3 solicited AE (Day 28): number analyzed (Participants) | 6
  PCS, Grade 3 solicited AE (Day 28) | -1.220 [-2.82 to 2.55]
  PCS, No Grade 3 solicited AE (Day 7): number analyzed (Participants) | 42
  PCS, No Grade 3 solicited AE (Day 7) | 0.000 [-11.19 to 13.58]
  PCS, No Grade 3 solicited AE (Day 21): number analyzed (Participants) | 42
  PCS, No Grade 3 solicited AE (Day 21) | 0.180 [-11.32 to 13.58]
  PCS, No Grade 3 solicited AE (Day 28): number analyzed (Participants) | 42
  PCS, No Grade 3 solicited AE (Day 28) | -0.130 [-6.36 to 13.58]
  MCS, Grade 3 solicited AE (Day 7): number analyzed (Participants) | 6
  MCS, Grade 3 solicited AE (Day 7) | -1.770 [-11.08 to 2.50]
  MCS, Grade 3 solicited AE (Day 21): number analyzed (Participants) | 6
  MCS, Grade 3 solicited AE (Day 21) | -0.565 [-2.35 to 2.47]
  MCS, Grade 3 solicited AE (Day 28): number analyzed (Participants) | 6
  MCS, Grade 3 solicited AE (Day 28) | 0.015 [-6.24 to 2.50]
  MCS, No Grade 3 solicited AE (Day 7): number analyzed (Participants) | 42
  MCS, No Grade 3 solicited AE (Day 7) | 0.480 [-10.43 to 11.83]
  MCS, No Grade 3 solicited AE (Day 21): number analyzed (Participants) | 42
  MCS, No Grade 3 solicited AE (Day 21) | 0.140 [-5.10 to 7.33]
  MCS, No Grade 3 solicited AE (Day 28): number analyzed (Participants) | 42
  MCS, No Grade 3 solicited AE (Day 28) | 0.000 [-7.29 to 11.83]

15. Secondary Outcome: Assessment of Changes From Baseline (Day 0) for Quality Adjusted Life Years (QALY) Weekly Scores for All Subjects Who Did and Who Did Not Report Any Grade 3 Solicited Symptoms Post Vaccination.
Description: Median and range of the change from baseline of the SF-36v2 score are presented for each time point. The assessed parameters for change from baseline were QALY scores. For all subscale component, scores range from 0 to 100, with high scores indicating high levels of functioning/quality of life. There was only 1 study participant > 64 years of age and that experienced no grade 3 solicited symptoms. Hence, weekly questionnaire was assessed only on the 18-64 age category subjects.
Time Frame: Day 0 (baseline) and at Days 7 and 21 QoL evaluation (post dose 1) and Day 28 QoL evaluation (post dose 2)
Population: Analysis were performed on the Total Vaccinated cohort (18-64 years of age) which included all vaccinated subjects within 18 to 64 years of age and for whom safety data were available. Only subjects with score test results were included.
Measure: Median (Full Range); unit: QALY scores
Arm/Group | Influenza A (H5N1) Virus Monovalent Vaccine 18-64 Years Group
Number analyzed (Participants) | 48
QALY scores
  QALY score, Grade 3, Day 7: number analyzed (Participants) | 5
  QALY score, Grade 3, Day 7 | 0.000 [-0.17 to 0.04]
  QALY score, Grade 3, Day 21: number analyzed (Participants) | 6
  QALY score, Grade 3, Day 21 | 0.021 [-0.17 to 0.07]
  QALY score, Grade 3, Day 28: number analyzed (Participants) | 6
  QALY score, Grade 3, Day 28 | -0.021 [-0.19 to 0.04]
  QALY score, No Grade 3, Day 7: number analyzed (Participants) | 42
  QALY score, No Grade 3, Day 7 | 0.000 [-0.25 to 0.33]
  QALY score, No Grade 3, Day 21: number analyzed (Participants) | 42
  QALY score, No Grade 3, Day 21 | 0.000 [-0.25 to 0.33]
  QALY score, No Grade 3, Day 28: number analyzed (Participants) | 41
  QALY score, No Grade 3, Day 28 | 0.000 [-0.16 to 0.33]

16. Secondary Outcome: Time Taken to Return to (or go Beyond) the Baseline (Day 0) Value in the SF-36v2 Daily Questionnaire Subscale Component, Summary Component and QALY Scores in Subjects Who Reported Unsolicited AEs Post Vaccination Dose 1
Description: The assessed parameters were Physical functioning (PF), Physical-health related role limitations (RP), Bodily pain (BP), General health (GH), Vitality (VT), Social functioning (SF), Emotional health related role limitations (RE), Mental health (MH) and physical and mental component summary measures (PCS, MCS) and QALY for subjects who reported unsolicited AEs in the first 7 days after Dose 1. Only negative deviations from baseline were considered. On any variable, if there was a negative deviation from baseline, then if and only if the value returned to baseline or above within the 7 days after dose 1, the number of days required to return to baseline or above was calculated. On any variable, if there was no variation within the 7 days after dose 1, then nothing was counted. If there was more than one negative deviation from baseline and more than one recovery, then only the first was considered. Analyses by age category were not performed for the daily SF-36v2 questionnaire results.
Time Frame: During the 7 days after Dose 1
Population: Analysis was performed on the Total Vaccinated cohort which included all vaccinated subjects who reported an unsolicited AE in the 7 days after Dose 1. Only subjects with negative deviations from baseline were analyzed.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Influenza A (H5N1) Virus Monovalent Vaccine Group
Number analyzed (Participants) | 29
Days
  PF: number analyzed (Participants) | 15
  PF | 1.6667 (0.8997)
  RP: number analyzed (Participants) | 11
  RP | 1.5455 (1.2136)
  BP | 1.7931 (0.9776)
  GH: number analyzed (Participants) | 19
  GH | 1.8947 (1.3289)
  VT: number analyzed (Participants) | 23
  VT | 1.6522 (1.1912)
  SF: number analyzed (Participants) | 11
  SF | 1.5455 (0.8202)
  RE: number analyzed (Participants) | 7
  RE | 1.5714 (1.1339)
  MH: number analyzed (Participants) | 15
  MH | 1.6000 (0.9103)
  PCS: number analyzed (Participants) | 26
  PCS | 2.1154 (1.3365)
  MCS: number analyzed (Participants) | 19
  MCS | 1.8947 (1.1970)
  QALY: number analyzed (Participants) | 25
  QALY | 1.8400 (1.2806)

17. Secondary Outcome: Quantitative Differences Between SF-36v2 Questionnaire Responses, and the Solicited Local and General Adverse Event Data Provided on Diary Cards
Description: The analysis of Quantitative differences between SF-36v2 questionnaire responses, and the solicited local and general adverse event data provided on diary cards was invalidated as the differences in scale between the measures could not be reconciled.
Time Frame: After the first and second vaccine doses
Population: The analysis of Quantitative differences between SF-36v2 questionnaire responses, and the solicited local and general adverse event data provided on diary cards was invalidated as the differences in scale between the measures could not be reconciled.
Arm/Group | Influenza A (H5N1) Virus Monovalent Vaccine Group
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Serious Adverse Events: From Day 0 up to Day 385; Solicited local and general symptoms: During the 7-day (Days 0-6) post-vaccination period after each vaccination; Unsolicited symptoms: During the 21-day (Day 0-20) post-vaccination period after each vaccination
Groups:
- Influenza A (H5N1)Virus Monovalent Vaccine ˃64 Years Group: Subjects ˃64 years of age received 2 doses of Influenza A (H5N1) Virus Monovalent Vaccine, Adjuvanted (A/Indonesia) at Days 0 and 21. The vaccine was administered intramuscularly in the deltoid of the non-dominant arm at Day 0 and dominant arm at Day 21.
Arm/Group | Influenza A (H5N1) Virus Monovalent Vaccine 18-64 Years Group | Influenza A (H5N1)Virus Monovalent Vaccine ˃64 Years Group
All-Cause Mortality (participants affected / at risk) | 0/49 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/49 | 0/1
Other Adverse Events (participants affected / at risk) | 46/49 | 1/1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Influenza A (H5N1) Virus Monovalent Vaccine 18-64 Years Group (N=49) | Influenza A (H5N1)Virus Monovalent Vaccine ˃64 Years Group (N=1)
Pain (General disorders) | 45 | 1
Redness (General disorders) | 6 | 0
Swelling (General disorders) | 7 | 0
Fatigue (General disorders) | 27 | 0
Gastrointestinal symptoms (General disorders) | 12 | 0
Headache (General disorders) | 20 | 0
Joint pain (General disorders) | 14 | 0
Muscle ache (General disorders) | 33 | 0
Shivering (General disorders) | 10 | 0
Sweating (General disorders) | 7 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.